CLINICAL TRIAL: NCT07288515
Title: Observational Prospective Study of Acalabrutinib in Chronic Lymphocytic Leukemia Therapy in Real Clinical Practice in Belarus.
Brief Title: Observ Prosp Study of Acalabrutinib in CLL Therapy in Real Clinical Practice in Belarus
Acronym: ALICIA(BY)
Status: Not yet recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D8220R00090
Record Dates: First submitted 2025-11-17; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with CLL: no control group or comparator involved

SUMMARY:
to address critical gap in knowledge, providing essential data on the real-world effectiveness, safety, associated with acalabrutinib treatment in patients with CLL

DETAILED DESCRIPTION:
This observational, prospective, multi-center study aims to gather real-world data (RWD) on acalabrutinib's use in routine clinical practice for CLL treatment in Belarus. Patients will be monitored without intervention, and all treatment decisions will be at the clinician's discretion. The study duration per patient will be approximately two years, with periodic data collection at regular intervals, ensuring comprehensive assessment of treatment effectiveness, patient safety, and quality of life metrics.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Confirmed diagnosis of CLL.
* Newly prescribed acalabrutinib monotherapy within the previous four weeks preceding study enrolment. Monotherapy is defined as acalabrutinib prescribes without concomitant administration (or planned initiation) of other anti-leukemic agents (e.g. obinutuzumab, venetoclax, bendamustine) within ± 30 days of acalabrutinib initiation.
* Treatment-naïve or R/R CLL.
* Ability and willingness to provide informed consent for study participation.

Exclusion Criteria:

* Patients not satisfying any of the inclusion criteria.
* Prior treatment with any BTK inhibitor.
* Participation in other ongoing clinical trials.
* Pregnant or breastfeeding females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises adult patients (≥18 years old) diagnosed with CLL, who have been newly prescribed acalabrutinib monotherapy within four weeks prior to study enrolment. This includes both treatment-naïve patients and patients with relapsed/refractory (R/R) CLL.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to treatment discontinuation | up to 25 months
  defined as the duration (in days) from the initiation of acalabrutinib therapy until the earliest of:
  1. documented permanent treatment discontinuation as recorded in the patient's medical chart, or
  2. death from any cause

SECONDARY OUTCOMES:
Reasons for treatment discontinuation | up to 25 months
  Collected from source medical documents (e.g., progression, toxicity, patient preference, physician's decision).
Rates for dose modifications | up to 25 months
  numerical count of dose reductions or holds, and categorization of underlying reasons (e.g., toxicity, drug interactions, comorbidities), derived from medical records
reasons for dose modifications | up to 25 months
  numerical count of dose reductions or holds, and categorization of underlying reasons (e.g., toxicity, drug interactions, comorbidities), derived from medical records
Subsequent treatments | up to 25 months
  qualitative categorical descriptions of therapies following acalabrutinib discontinuation
Treatment interruptions | up to 25 months
  temporary discontinuation of acalabrutinib lasting ≥7 days but <30 days, with documented intent to resume treatment. Interruptions and their documented reasons will be captured from medical records

OTHER OUTCOMES:
PFS measures, including one- and two-year rates | up to 25 months
  PFS, defined as the time from first dose to documented progression or death, assessed by Investigator based on clinical evaluations and diagnostic imaging, when available.
OS rates | up to 25 months
  OS rates at one and two years of follow-up defined as proportion of alive participants at the given timepoint

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: ICF, CSR
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/